CLINICAL TRIAL: NCT03543618
Title: Evaluation of Dental Implant Placement in the Sloped Alveolar Ridge
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201704081DIPC
Record Dates: First submitted 2018-03-20; First posted 2018-06-01 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2017-10

CONDITIONS: Atrophy of Edentulous Alveolar Ridge
Keywords: dental implant; edentulous ridge

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Sham Comparator): Installation of conventional design dental implant
  Interventions: Device: Control
- Sloped (Active Comparator): Installation of sloped design dental implant
  Interventions: Device: Sloped

INTERVENTIONS:
Device: Sloped — Placement of implant with sloped design
  Other Names: "Astra" OsseoSpeedTM Profile EV
  Arms: Sloped
Device: Control — Placement of implant with conventional design
  Other Names: "Astra" OsseoSpeedTM EV
  Arms: Control

SUMMARY:
The aim of this study was to investigate the therapeutic effect of sloped dental implants. It can reduce the need of osteoectomy, reduce discomfort of procedures, and is easier for maintenance.

DETAILED DESCRIPTION:
20 OsseoSpeed ™ Profile EV and 20 OsseoSpeed ™ EV groups will be randomly implanted into the oblique edentulous ridges of subjects, and the treatment response will be monitored for 3 years. The implantation area will be randomly divided into two groups, One group was treated with OsseoSpeed ™ Profile EV (sloped group) and the other group was treated with OsseoSpeed ™ EV (control group). The same patient had the same implant as the same quadrant.

The patient will be followed up regularly for follow-up, followed by clinical attachment level, probing depth, bleeding on probing, keratinized gingival width (Keratinized gingiva), mobility (mobility) and other clinical indicators of the measurement, regular dental radiography, gingival crevicular fluid (GCF) collection and bone integration measurement.

After six months of implantation, prosthesis will delivered and loaded functionally, and regular follow-up will be arranged. In each time of follow-up, examination will be carried out with regards to periodontal pocket depth, clinical attachment height, periodontal bleeding index, keratinized gingival width, and other clinical indicators of the measurement, at the end of the experiment, that is, after three years, and then a dental root film irradiation, GCF collection and osseointegration measurement.

ELIGIBILITY:
20-80 years old with appropriate oral cleaning ability; the computer tomography shows > 1 mm buccolingual discrepancy of alveolar ridge height; no generalized periodontitis, or had history of periodontitis but has been completed treatment; no major systemic infection or major systemic illness; not taken antibiotics in the past two weeks Not pregnant or breastfeeding

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-03-15 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Clinical assessment of the status of osseointegration | up to 3 years
  radiographic bone level, bone consolidation index (ISQ)

SECONDARY OUTCOMES:
The health status of adjacent teeth | 0 day, 6 months, 1 year, 2 years, 3 years
  radiographic bone level, clinical attachment level, pocket depth, periodontal bleeding (bleeding on probing), keratinized gingival width (masticatory mucosa width)
The peri-implant health | 1 year, 2 years, 3 years
  radiographic bone level, clinical attachment level, pocket depth, periodontal bleeding (bleeding on probing), keratinized gingival width (masticatory mucosa width)
Biomarkers in the gingival crevicular fluid of adjacent teeth | 0 day, 6 months, 1 year, 2 years, 3 years
  Inflammatory markers such as Interleukin-1 beta, matrix metalloproteinase-8, Interleukin-8, or Interleukin-10
Biomarkers in the gingival crevicular fluid of dental implant | 1 year, 2 years, 3 years
  Inflammatory markers such as Interleukin-1 beta, matrix metalloproteinase-8, Interleukin-8, or Interleukin-10

CONTACTS AND LOCATIONS:
Overall Officials: Po-Chun Chang, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan